CLINICAL TRIAL: NCT00929604
Title: Effectiveness of HIV Viral Load Monitoring of Patient Outcome in Resource-Poor Settings
Brief Title: HIV Viral Load Monitoring in Resource-Poor Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Adult AIDS Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VLS
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: HIV; AIDS; HIV Infections
Keywords: HIV; AIDS; Zambia; viral load; antiretroviral therapy; cluster randomization; ART monitoring; treatment failure; randomized clinical trial; treatment naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (No Intervention): Standard of care arm: utilizes the current standard of care per Zambian national guidelines to determine treatment failure and eligibility for second-line ART. HIV-1 viral load measurement is performed if the criteria for either immunologic (i.e., CD4+ lymphocyte count-based) or clinical treatment failure are fulfilled. If both immunologic and clinical treatment failure criteria are fulfilled, the ART regimen is changed to second-line without VL testing.
- Routine HIV-1 viral load testing (Experimental): Routine viral load testing arm: Routine HIV viral load testing at ART initiation (baseline) and at 3, 6, 12, 18, 24, 30 and 36 months thereafter.
  Interventions: Other: HIV-1 viral load testing

INTERVENTIONS:
Other: HIV-1 viral load testing — Plasma HIV-1 RNA viral load testing performed at ART initiation (baseline) and at 3, 6, 12, 18, 24, 30, and 36 months thereafter. Routine viral load results are provided to clinicians for the management of the participant's HIV treatment.
  Other Names: Viral load measured by the Roche Amplicor HIV-1 RNA Monitor kit (version 1.5; Roche Molecular Diagnostics, Pleasanton, CA, USA).
  Arms: Routine HIV-1 viral load testing

SUMMARY:
No randomized clinical trial to date has demonstrated a survival benefit of using regular HIV-1 ribonucleic acid (RNA) viral load (VL) testing to monitor patients' responses to antiretroviral therapy (ART) for HIV infection. The measurement of VL is recommended to monitor the response to ART in developed countries. In resource-constrained settings, the World Health Organization (WHO) does not recommend routine VL testing, in part due to the cost and complex infrastructure needed for reliable results. In these settings, WHO has proposed the use of clinical and CD4+ lymphocyte-based criteria to guide treatment decisions. However, multiple studies have demonstrated the poor performance of these criteria in sub-Saharan Africa and the frequent discordance between immunologic and virologic responses to ART.

The use of routine viral load monitoring should be evaluated in resource-constrained settings. The investigators hypothesize that routine viral load testing of patients on ART will improve patient survival, decrease disease progression and development of drug resistance, and will be feasible and cost-effective for resource-constrained settings.

DETAILED DESCRIPTION:
The study 'Effectiveness of HIV Viral Load Monitoring on Patient Outcome in Resource-Poor Settings,' is a dual-arm, cluster randomized trial to evaluate the use of routine plasma HIV-1 VL monitoring to improve survival and decrease HIV disease progression in patients receiving ART. The primary objective is to assess mortality at 36 months among ART naïve patients initiating therapy and receiving care at facilities with access to routine HIV VL testing (at ART initiation, at 3 months and at every 6 months thereafter) compared to those initiating first regimens and receiving care at facilities according to our local standard of care (which uses immunological [i.e. CD4+ lymphocyte count-based]and clinical criteria to diagnose treatment failure, with discretionary VL testing when the two do not agree).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection (according to local standard rapid testing algorithms)
* Age 18 years or greater
* Able and willing to provide informed consent to participate
* Eligible for antiretroviral therapy per Zambian national guidelines, which are any of the following:

  * CD4+ cell count less than 200 cells/mm3;
  * WHO Stage IV disease; or
  * WHO Stage III disease and CD4+ cell count less than 350 cells/mm3
* Residence in the geographical catchment area of the VLS clinic and intent to remain there for the duration of the study
* Willingness to adhere to the study visit schedule and to be followed-up at home in the event of a missed study visit
* Initiating ART on the day of VLS enrollment, informed consent, and baseline blood collection

Exclusion Criteria:

* Receipt of more than 7 days (cumulative) of prior antiretroviral therapy at any time prior to study entry, with the exception of zidovudine and/or single dose nevirapine for prevention of mother-to-child transmission;
* Any exposure to antiretroviral therapy in the past one month
* A condition that, in the opinion of the investigators, would interfere with adherence to study requirements (e.g., mental illness or active drug or alcohol use or dependence)
* Serious illness requiring referral to hospital at the time of ART initiation
* For patients seeking care at sites randomized to the standard of care arm: participation in another research protocol that offers routine viral load testing
* Unwillingness to consent to all aspects of study protocol including blood specimen storage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2112 (Actual)
Dates: Start 2006-12; Primary Completion 2012-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Patient survival | 36 months

SECONDARY OUTCOMES:
To assess HIV clinical disease progression (weight, CD4 cell response, incident opportunistic infections) | 36 months
To assess the impact of more rapid ART regimen switching on available second and third-line treatment options | 36 months
To monitor the effectiveness of newer antiretroviral medications introduced in Zambia (principally tenofovir) | 36 months
To characterize the timing and sequence of HIV drug resistance development among patients in each study arm | 36 months
To assess the feasibility, acceptability, and cost effectiveness of the two management strategies in a resource-constrained sub-Saharan African setting | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Saag, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

REFERENCES:
- [Derived] Koethe JR, Westfall AO, Luhanga DK, Clark GM, Goldman JD, Mulenga PL, Cantrell RA, Chi BH, Zulu I, Saag MS, Stringer JS. A cluster randomized trial of routine HIV-1 viral load monitoring in Zambia: study design, implementation, and baseline cohort characteristics. PLoS One. 2010 Mar 12;5(3):e9680. doi: 10.1371/journal.pone.0009680. PMID 20300631